CLINICAL TRIAL: NCT03685669
Title: Detection of Early-stage Lung Cancer by Using Methylation Signatures in Circulating Tumor DNA
Brief Title: Non-Invasive ctDNA Methylation Detection for Lung Nodule Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Singlera Genomics Inc. (Industry)
Responsible Party: Principal Investigator, Lu Shun, Principle Investigator, Shanghai Chest Hospital
Other Study IDs: KS1811
Record Dates: First submitted 2018-09-10; First posted 2018-09-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-09

CONDITIONS: Lung Nodule
Keywords: DNA methylation; ctDNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung nodule group
- Healthy Control group

SUMMARY:
Low-dose computed tomography (LDCT) is recommended for early-stage lung cancer screening. However, it is often difficult to determine indolent lesions from more aggressive tumors without an invasive intervention or prolonged follow-up period. Thus, the main purpose of this study is to develop a non-invasive method to detect lung-cancer specific circulating tumor DNA (ctDNA) in blood, which can greatly improve the specificity of lung cancer early screening.

DETAILED DESCRIPTION:
In this study, the investigators sought to explore sensitive and specific methylation biomarkers that are highly prevalent in lung cancer. It is the first time to perform screening assay on healthy, lung nodule, and lung cancer tissues to identify preliminary set of highly prevalent methylation markers, and then refined these markers by removing regions were unstable in matched plasma samples. Next, investigators interrogated significant methylation marker regions enriched in lung nodules of training sample set to buildup a non-invasive biomarker classification model to discriminate cancerous nodules from benign lesions. Eventually, the model in patient lung nodule samples were validated.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or above with pulmonary nodule(s) found by LDCT, mean diameter below 30mm.
2. The nodule lesion is peripheral, no signs of lymphatic infiltration or distal metastasis.
3. Fit and consent to surgical resection.
4. Agree to participate in this study and sign informed consents.

Exclusion Criteria:

1. Fail to understand or agree to sign informed consent.
2. Patients who did not follow the test plan for timely blood collection or did not cooperate with the study follow-up work.
3. Patients with previous history of cancer and/or cancer treatment such as surgery, radiotherapy, chemotherapy or targeted therapy.
4. Failing to meet the requirements for blood sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who have single or multiple lung nodules detected by LDCT and are about to undergo surgery; healthy sex and age matched controls
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Noninvasive assisted diagnosis of benign and malignant pulmonary nodules | 1 year
  The biomarker classification model can be used to differentiate patients, who had positive LDCT results, with benign or malignant lung nodules.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No